# TRIAL TO ASSESS THE EFFICACY OF LENVATINIB IN METASTATIC NEUROENDOCRINE TUMORS (TALENT STUDY)

| Sponsor: | GETNE (Grupo Español de Tumores Neuroendrocrinos) |
|-----------------|---------------------------------------------------|
| Author: | Silvia Lladosa Marco |
| Document type: | Statistical Analysis Plan |
| Eudract number: | 2015-001467-39 |
| Phase: | II |
| Version: | 2.0 |
| Release date: | 04/JUN/2020 |

**Notice:** Part or all the information included in this document may be unpublished material and it should be treated as <u>confidential and property of the sponsor</u>. It may not be disclosed to any unauthorized person, including publications and presentations, without the written consent of the Sponsor.

 Date: June 04, 2020

## SIGNATURE PAGE FOR THE STATISTICAL ANALYSIS PLAN

# TRIAL TO ASSESS THE EFFICACY OF LENVATINIB IN METASTATIC NEUROENDOCRINE TUMORS (TALENT STUDY)

| Sponsor: | GETNE (Grupo Español de Tumores Neuroendrocrinos) |
|---|---|
| Author: | Silvia Lladosa Marco |
| Sponsor contact person: | Dr. Jaume Capdevila |
| Sponsor, signature and date: | 10/6/20 |
| Author, signature and date: | [2] 12/06/2020 |

## 1. Synopsis

| Type of application | |
|---|---|
| Sponsor | GETNE (Grupo Español de Tumores Neuroendrocrinos) París 162, Pral. 1ª. 08036, Barcelona Phone:93 451 17 24; Fax: 93 451 43 66 |
| Clinical trial title | "TRIAL TO ASSESS THE EFFICACY OF LENVATINIB IN METASTATIC NEUROENDOCRINE TUMORS (TALENT STUDY)." |
| Protocol number | GETNE1509 (TALENT) |
| Study Coordinator and Principal Investigator | Dr. Jaume Capdevila Medical Oncology Department. Gastrointestinal and Endocrine Tumor Unit Vall d'Hebron University Hospital Pg Vall d'Hebron, 119-129; 08035 Barcelona Tel. +34934894350; Fax. +34932746781 jacapdevila@vhebron.net; jcapdevila@onco.cat |
| Expected sites | Approximately 25 sites in several countries in Europe (planned sites in Spain, Italy, United Kingdom and Austria) |
| Central Ethics Committee/Institutional Review Board | <ul> <li>CEIC Hospital Universitari Vall d'Hebron</li> <li>CEIC Área 4 – Hospital Universitario Ramón y Cajal</li> <li>CEIC Área 5 – Hospital Universitario La Paz</li> <li>CEIC Área 11 – Hospital 12 de Octubre</li> <li>Comité Ético de Investigación Clínica de Asturias</li> <li>Comité Ético de Investigación Clínica de Cantabria</li> <li>CEIC Hospital Universitari de Bellvitge</li> <li>CEIC Euskadi</li> <li>CEIC de los Hospitales Universitarios Virgen Macarena – Virgen del Rocío de Sevilla</li> </ul> |
| Name and qualification of the persons in charge of Monitoring | Experior, S.L. C/ Vicente Galmés, 1A; 46139 La Pobla de Farnals (Valencia) |

| ALENT Statistical Analysis Plan | version 2.0 Date: June 04, 2020 |
|---|---|
| | Tel.: 902.105.255; Fax: 96.145.21.91 |
| Investigational drug | Lenvatinib |
| | Lenvatinib will be provided as 4-size hydroxypropyl methylcellulose (HPMC) capsules in 2 strengths differentiated by color: 4-mg capsule (yellowish-red cap and body) and 10-mg capsule (yellowish-red cap with yellow body). Dosing schedule of 24 mg once a day (two 10-mg capsules + one 4-mg capsule) has been selected for continued lenvatinib |
| | development. |
| Trial phase | II |
| Objectives | Primary objective To assess the efficacy of lenvatinib on tumor objective response rate in two independent cohorts of patients with advanced neuroendocrine tumors: patients with advanced/metastatic G1/G2 pancreatic neuroendocrine tumors after progression to a previous targeted agent (cohort A), and patients with advanced/metastatic G1/G2 neuroendocrine tumors of gastrointestinal tract after failure to somatostatin analogues therapy (cohort B). Secondary objectives To determine the safety and tolerability of lenvatinib. To estimate the early tumor shrinkage rate and the deepness of response of lenvatinib in each cohort of patients. To estimate progression-free survival in both cohorts of patients. Exploratory objectives To evaluate biochemical response (changes in CgA and NSE levels) and its association with response rate and progression-free survival. To assess whether baseline tumor and blood biomarkers may be predictive of response to lenvatinib. To explore additional hypotheses related to biomarkers and relationship to lenvatinib, neuroendocrine tumors, other |

 Date: June 04, 2020

| TALENT Statistical Analysis Plan | Version 2.0 Date: June 04, 2020 |
|---|---|
| | endocrine disorders and/or cancer which may arise from internal or external research activities. |
| Design | Prospective, international, multi-center, open label, stratified, exploratory phase II study evaluating the efficacy and safety of lenvatinib. |
| Primary endpoint | The primary endpoint of the study is overall response rate (ORR) by RECIST v 1.1 upon central radiologic assessment. |
| Study population and total number of subjects | Patients with advanced/metastatic, histologically confirmed, grade 1/2 (G1/G2) of 2010 WHO classification neuroendocrine tumors of the pancreas after progression to a previous targeted agent (cohort A) or gastrointestinal tract after progression to somatostatin analogues (cohort B). Number of patients: 110 patients in total (55 per each cohort). |
| Approximate duration of subject participation | 24 months |
| Calendar and estimated completion dates | Recruitment Start: September 2015 End of Recruitment Period: March 2017 3rd Tumor assessment of LP (Primary Analysis): July 2017 Database Lock for Interim Analysis: October 2017 End of Follow up Period: March 2019 FPFV: September 2015 LPLV: September 2018 Clinical Study Report: September 2019 |

| 2. Tab | ple of contents | |
|---|---|---|
| 1. Sy | nopsis | 3 |
| 2. Tal | ble of contents | 6 |
| 3. Ab | breviations | 7 |
| 4. Stu | ıdy objectives and variables | 8 |
| 4.1 | Primary objective(s) and primary variable(s) | |
| 4.2 | Secondary objective(s) and secondary variables | |
| | secondary objectives are: | |
| 4.3 | Exploratory objective(s) and variables | |
| The e | exploratory objectives are: | |
| | pratory variables: | |
| 5. Stu | ıdy populations | 10 |
| | itistical strategy | |
| 6.1 | Primary analysis | |
| 6.1.1 | Summary statistics | |
| 6.1.2 | Statistical inference | |
| 6.2 | Secondary analysis | |
| | secondary analysis will be based on the Full Analysis Set and the Safety Ana | |
| Set | | 11 |
| 6.2.1 | Summary statistics | 11 |
| 6.2.2 | Statistical inference | 12 |
| 6.3 | Exploratory analysis | 12 |
| 6.4 | Subgroup analysis | |
| 6.5 | Safety analysis | _ |
| 6.5.1 | Summary statistics | |
| 6.5.2 | Statistical inference | |
| 6.6 | Demographic and baseline characteristics | |
| 6.7 | Concomitant medications | |
| 6.8 | Statistical significance level | |
| 6.9 | Statistical model assumptions | |
| 6.10<br>6.11 | Transformation of expected variables Handling of missing data | |
| 6.12 | Description of the softwares to be used for data analysis | |
| 6.13 | Interim analysis protocol | |
| | ferences | |
| i. Re | C C C C C C C C C C C C C | 16 |

Confidential Version 2.0

GETNE
TALENT Statistical Analysis Plan

 Date: June 04, 2020

#### 3. Abbreviations

AE:

Adverse Event

CgA:

Chromogranin A

CR:

Complete Response

DpR:

Deepness of Response

ECG:

Electrocardiogram

eCRF:

electronic Case Report Form

ETS:

Early Tumor Shrinkage

G1:

Grade 1

G2:

Grade 2

**GETNE:** 

Grupo Español de Tumores Neuroendrocrinos

HPMC:

Hydroxypropyl Methylcellulose

NSE:

Neuron Specific Enolase

OOR:

Objective Response Rate

OS:

**Overall Survival** 

PFS:

Progression-Free Survival

PI:

Principal Investigator

PR:

Partial Response

RECIST:

Response Evaluation Criteria In Solid Tumors

SAE:

Serious Adverse Event

WHO:

World Health Organization

## 4. Study objectives and variables

## 4.1 Primary objective(s) and primary variable(s)

To assess the efficacy of lenvatinib on tumor objective response rate (ORR), complete (CR) and partial responses (PR) in two independent cohorts of patients with advanced/metastatic G1/G2 neuroendocrine tumors: patients with pancreatic neuroendocrine tumors after progression to a previous targeted agent (cohort A), and patients with neuroendocrine tumors of the gastrointestinal tract after failure to somatostatin analogues therapy (cohort B).

The ORR is defined as the proportion of subjects who have best overall response of CR or PR (by RECIST criteria):

$$ORR = \frac{CR + PR}{Total \ of \ patients}$$

## 4.2 Secondary objective(s) and secondary variables

The secondary objectives are:

- To determine the safety and tolerability of lenvatinib.
- To estimate the early tumor shrinkage rate and the deepness of response of lenvatinib in each cohort of patients.
- To estimate progression-free survival in both cohorts of patients.

#### Secondary variables:

- To determine the safety and tolerability of lenvatinib. Safety will be assessed by adverse events (AEs) and serious adverse events (SAEs). Echocardiogram results (LVEF reductions) and QTc (using the QTcB and QTcF values) prolongations will be examined. QTc prolongation will be examined through the adverse events.
- To estimate the early tumor shrinkage (ETS) rate and the deepness of response
   (DpR) of lenvatinib in each cohort of patients:
  - ETS rate is defined as 20% reduction in target lesions after the first 6 weeks of treatment (first tumor assessment).
  - DpR is defined as percentage of maximum tumor shrinkage observed at the nadir (minimum value of total sum of diameters) compared with baseline.

To assess ETS and DpR, total sum of diameters obtained in all tumor assessments will be considered.

• To estimate progression-free survival (PFS) in both cohorts of patients. PFS is defined as the time from the date of treatment start (C1D1) to the date of first documentation of disease progression or death (whichever occurs first) using RECIST 1.1.

 Date: June 04, 2020

To evaluate PFS, it will be considered:

- Start date of study drug
- o Progression disease date or death date (whichever comes first)

PFS censoring rules will follow FDA guidance in 2007 [1]:

Table A. PFS 1 (includes documented progression only)

| Situation | Date of Progression or Censoring | Outcome |
|---|---|---|
| No baseline tumor assessments | Randomization | Censored |
| Progression documented between scheduled | Earliest of: | Progressed |
| visits | <ul> <li>Date of radiological assessment showing new lesion (if progression is based on new lesion); or</li> <li>Date of last radiological assessment of measured lesions (if progression is based on</li> </ul> | |
| | increase in sum of measured lesions) | 6 1 |
| No progression | Date of last radiological assessment of measured lesions | Censored |
| Treatment discontinuation for undocumented progression | Date of last radiological assessment of measured lesions | Censored |
| Treatment discontinuation for toxicity or other reason | Date of last radiological assessment of measured lesions | Censored |
| New anticancer treatment started | Date of last radiological assessment of measured lesions | Censored |
| Death before first PD assessment | Date of death | Progressed |
| Death between adequate assessment visits | Date of death | Progressed |
| Death or progression after more than one missed visit | Date of last radiological assessment of measured lesions | Censored |

## 4.3 Exploratory objective(s) and variables

The exploratory objectives are:

- To evaluate biochemical response (changes in CgA, 5-HIAA and NSE levels) and its association with response rate and progression-free survival.
- To assess whether baseline tumor and blood biomarkers may be predictive of response to lenvatinib.
- To explore additional hypotheses related to biomarkers and relationship to lenvatinib, neuroendocrine tumors, other endocrine disorders and/or cancer which may arise from internal or external research activities.

#### **Exploratory variables:**

- The changes in tumor markers (CgA, 5-HIIAA and NSE) will be analysed by cohort and significant reductions defined as 50% reduction or more regarding the baseline values will be calculated.
- The relationship between reductions and PFS and radiological response will be assessed.

EudraCT number: 2015-001467-39

Confidential Version 2.0

 Date: June 04, 2020

The second and third exploratory objectives will be assessed in the final analysis not in the interim analysis. According to the biomarkers that are available, the analysis of these objectives will be specified.

## 5. Study populations

The analysis sets will be defined as follows:

- <u>Full Analysis Set</u> will include all allocated subjects. This will be primary analysis set for the efficacy endpoints.
- Per Protocol Analysis Set will include those subjects who were allocated and received at least one dose of the assigned study drug and had no major protocol deviations. The subjects will complete both baseline and at least one post-baseline tumor assessments (week 6). Experior will send a list of major protocol deviations to establish the per-protocol set after the close out of data base. The PI (Dr. Capdevila) will decide which patients should be excluded to define the per protocol analysis set.
- <u>Safety Analysis Set</u> will include all subjects who were allocated and received at least one dose of the study drug and had at least one post-baseline safety evaluation (week 6). This will be the analysis set for all safety evaluations.

## 6. Statistical strategy

Below are detailed the statistical aspects of the data analysis.

#### 6.1 Primary analysis

All efficacy analyses will be based primarily on the Full Analysis Set and secondarily on the Per Protocol Analysis Set.

#### 6.1.1 Summary statistics

The ORR will be calculated by RECIST v1.1 upon central radiologic assessment, independently for each cohort.

Waterfall plots (2D and 3D) will be calculated to examine the changes in tumor lesions from baseline.

## 6.1.2 Statistical inference

It is not planned statistical inference.

 Date: June 04, 2020

## 6.2 Secondary analysis

The secondary analysis will be based on the Full Analysis Set and the Safety Analysis Set.

#### 6.2.1 Summary statistics

Secondary endpoints will be summarized with descriptive statistics. Continuous variables will be summarized with n, NA, mean, standard deviation, median and range. Frequency counts and percentage of subjects within each category will be provided for categorical data.

#### First secondary objective:

Safety analyses will be based on the Safety Analysis Set. All safety analyses will be summarized separately by cohort.

Adverse events will be classified into standardized medical terminology from the verbatim description (investigator term) using the Medical Dictionary for Regulatory Activities (MedDRA). Adverse events will be presented by preferred term (PT) and by system organ class (SOC).

Echocardiogram results (LVEF), and their changes from baseline will be summarized using descriptive statistics. Prolongation of QTc will be analysed using descriptive statistics and frequency tables.

The degree of exposure (dose, duration of treatment, interruptions/reductions of dose) will be assessed to determine the degree to which study safety can be assessed. These results will be presented with descriptive statistics (n, NA, mean, standard deviation, median and range).

#### Second secondary objective:

The ETS and DpR will be calculated for each cohort. Both ratios will be calculated using the total sum of diameters provided in tumor assessments by central radiology review.

#### Third secondary objective:

PFS will be calculated using start date of study drug and progression disease or death date (whichever occurs first), based on the Full Analysis set and Per-protocol Analysis Set. PFS censoring rules will follow FDA guidance in 2007 (see Table A).

OS will be calculated using start date of study (C1D1).

A Kaplan Meier survival analysis will be carried out to analyse PFS, providing the median and the corresponding 95% CI of time to progression. Survival curves will be reported.

#### 6.2.2 Statistical inference

Comparisons using log rank test or model of Cox proportional hazards multivariate analysis will be used if needed.

## 6.3 Exploratory analysis

## First secondary objective:

Significant reductions of tumor markers (CgA, 5-HIAA and NSE), defined as reductions of 50% or more regard the baseline values, will be showed by frequency tables.

To examine the relationship of biochemical response with PFS and radiological response the Kaplan-Meier and Chi-square/Fisher methods will be used.

## 6.4 Subgroup analysis

Subgroup analysis for ORR, PFS, OS, biochemical response (tumor markers) will be performed outside the indications of the study protocol. The following variables will be part of this analysis to explore differences between subgroups of subjects:

#### ORR:

- Origin of gastrointestinal NET.
- Functionality.
- Tumor burden (this information will be extract from central radiologic assessment).
- Number of previous lines (1, 2 or 3 lines) (only in pancreatic NET cohort).
- Concomitant use of somatostatin analogues.
- Previous treatment with everolimus or sunitinib (only in pancreatic NET cohort).

#### PFS:

- Origin of gastrointestinal NET.
- Tumor burden.
- Number of previous lines (1, 2 or 3 lines) (only in pancreatic NET cohort).
- Concomitant use of somatostatin analogues.


Date: June 04, 2020

-  Date: June 04, 2020
- Previous treatment with everolimus or sunitinib (only in pancreatic NET cohort).
- o ECOG.
- Prior surgery.
- Age (≤ 65 vs > 65 years).
- o Differentiation grade (G1/G2).
- Radiological response (upon central radiologic assessment).
- OS:
  - Functionality.
  - o Tumor burden.
  - Concomitant use of somatostatin analogues.

Survival curves will be calculated for OS

In addition to the subgroup analysis, it will be calculated:

- Duration of response will be assessed and represented graphically. It will be calculated as time since treatment initiation to progression disease.
- Time to follow-up will be described.

## 6.5 Safety analysis

The safety analysis has been included in secondary objective (see 6.2).

## 6.5.1 Summary statistics

Not applicable.

## 6.5.2 Statistical inference

Not applicable.

## 6.6 Demographic and baseline characteristics

Demographic and other baseline characteristics will be summarized and listed. For continuous demographic/baseline variables, results will be summarized and presented as n, number of not available data (NA), mean, standard deviation, median, and minimum and maximum values. For categorical variables, the number and percentage of subjects will be used.

 Date: June 04, 2020

Demographic and baseline characteristics variables are:

- Age
- Gender
- Menopausal status
- Race/ethnicity
- ECOG performance status
- TNM staging (tumor, nodules and metastasis)
- Time from diagnosis date to informed consent signature
- Time from metastatic diagnosis date to informed consent signature
- Histological characteristics: Differentiation grade, Ki67 expression, Miotic count, NYHA classification
- Medical and surgical history
- Previous anti-cancer treatments
- Functionality
- Origin of gastrointestinal NET

#### 6.7 Concomitant medications

Concomitant medications associated with an AEs will be coded to the appropriate Anatomical-Therapeutic-Chemical (ATC) code indicating anatomical main group and therapeutic subgroup.

## 6.8 Statistical significance level

A significance level of 5% will be considered.

 Date: June 04, 2020

## 6.9 Statistical model assumptions

The following assumptions will be verifying to guarantee t Student test (if applicable)

- Normality of data
- Variance homogeneity
- Independence in data

In case of applying a Cox regression model, proportional hazards assumption (graphically) will be checked.

## 6.10 Transformation of expected variables

• The ORR is defined as the proportion of subjects who have best overall response of CR or PR (by RECIST 1.1):

- The time to progression is defined as the difference between start of drug (C1D1) and the progression date or death (whichever occurs first) or the last tumor assessment documented.
- ETS rate is defined as 20% reduction in target lesions after the first 6 weeks of treatment.
- DpR is defined as percentage of maximum tumor shrinkage observed at the nadir (the minimum of total sum of diameters) compared with baseline.
- Overall survival is defined as the time from the start of drug (C1D1) to death.

## 6.11 Handling of missing data

No planned procedure of imputation of missing values. The analysis will be performed with the available data.

#### 6.12 Description of the softwares to be used for data analysis

Statistical programming and analyses will be performed using R [2] statistical software.

#### 6.13 Interim analysis protocol

The interim analysis will be performed when the last patient included in the corresponding cohort of the study will have at least two tumor assessments (12 weeks after the last patient recruited).

 Date: June 04, 2020

## 7. References

- 1. Guidance for Industry: Clinical Trail Endpoints the Approval of Cancer Drugs and Biologics (May 2007).
- 2. R Core Team (2015). R: A language and environment for statistical computing. R Foundation for Statistical Computing, Vienna, Austria. URL (http://www.R-project.org/).